CLINICAL TRIAL: NCT06242067
Title: Irinotecan in Combination With Trifluridine-tipiracil and Bevacizumab in Pre-treated Metastatic Colorectal Cancer
Brief Title: Second-line Treatment of Metastatic Colorectal Cancer
Acronym: BEV-TASIRI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: The Affiliated Hospital of Qingdao University (Other); Shandong Provincial Hospital (Other Government); Qianfoshan Hospital (Other); Binzhou People's Hospital (Other); Binzhou Medical University (Other); Yantai Yuhuangding Hospital (Other); Linyi Tumour Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KYLL-202210-057-1
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: colorectal cancer; bevacizumab; trifluridine-tipiracil/TAS-102; irinotecan
MeSH Terms: conditions — Colorectal Neoplasms | interventions — trifluridine tipiracil drug combination; Irinotecan; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Irinotecan,Trifluridine-tipiracil in combination with Bevacizumab (Experimental)
  Interventions: Drug: Trifluridine/tipiracil

INTERVENTIONS:
Drug: Trifluridine/tipiracil — patients received biweekly Trifluridine/tipiracil (30 mg/m2 twice daily; days 1-5), irinotecan (150 mg/m2; day 1) and bevacizumab (5 mg/kg; day 1).
  Other Names: Irinotecan; Bevacizumab

SUMMARY:
The goal of this multicenter, single-arm, observational cohort study is to investigate the efficacy and safety of irinotecan in combination with trifluridine-tipiracil and bevacizumab in colorectal cancer with prior oxaliplatin and fluoropyrimidine-based chemotherapy (including 5-FU/capecitabine/S-1) exposure in the metastatic setting or within 12 months of recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects are required to sign an informed consent form before starting the study-related procedure
2. Age 18-75 years old, male or female.
3. have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1, life expectancy >3 months.
4. Histologically or cytological proven metastatic or recurrent adenocarcinoma of the colon or rectum.
5. Prior treatment with a fluoropyrimidine (5-fluorouracil [5-FU] or capecitabine) and oxaliplatin with bevacizumab or cetuximab targeted therapy as the first-line regimen.
6. Recurrence or metastasis within 12 months after completion of adjuvant/neoadjuvant therapy with oxaliplatin and fluoropyrimidine-based drugs is also considered as the failure of first-line chemotherapy.
7. At least one measurable metastatic lesion, as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
8. Adequate organ function: bone marrow, kidney, liver function (within 7 days before treatment start) Absolute neutrophil count ≥ 1.5×109/L Platelet count ≥ 100×109/L Hemoglobin≥ 90g/L (no history of blood transfusion within 7 days); Creatinine clearance≥ 60 ml/min (Cockcroft-Gault formula) Bilirubin ≤ 1.5 x the upper limit of normal (ULN) Glutamate aminotransferase (AST)/ alanine aminotransferase (ALT) levels ≤2.5 x ULN or =< 5 x ULN if with hepatic metastases; Alkaline phosphatase (AKP) ≤ 2.5 x ULN or =< 5 x ULN if with hepatic metastases;
9. Urine protein <1+ or 24-hour urine protein <1 gram;
10. International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 x ULN or within the range if receiving anticoagulant therapy;
11. Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence; IUDs, etc) during the study period and within 90 days of the last study medication. All female patients will be considered fertile unless they have spontaneous menopause, artificial menopause, or sterilization (e.g., hysterectomy, bilateral adnexectomy, or radiation ovarian irradiation).

Exclusion Criteria:

1. First-line treatment with irinotecan;
2. Patients with KRAS/NRAS/BRAF wild-type and not treated with cetuximab in the first line.
3. Patients with dMMR/MSI-H (deficient mismatch repair/microsatellite instability-high) status;
4. Symptomatic brain or meningeal metastases (except for brain metastases that have undergone local radiotherapy or surgery for more than 6 months and stable disease control)
5. Previous or current severe bleeding (bleeding >30ml within 3 months), coughing up blood (>5ml of fresh blood within 4 weeks) or cerebrovascular accident (excluding lacunar cerebral infarction, minor cerebral ischemia or transient ischemic attack, etc.) within half a year before the first use of the study drug, myocardial infarction, unstable angina, poorly controlled arrhythmias (including QTc interval ≥450 ms for men and 470 ms for women≥) (QTc interval is calculated by Fridericia formula). According to the New York College of Cardiology (NYHA) standard class III or IV cardiac insufficiency or cardiac ultrasound: left ventricular ejection fraction (LVEF) < 50%.
6. Uncontrolled hypertension: systolic blood pressure >140mmHg, diastolic blood pressure > >90mmHg;
7. Digestive tract diseases or states that the investigator determines may affect drug absorption, including but not limited to active gastric and duodenal ulcers, ulcerative colitis and other digestive tract diseases or active bleeding in unresected gastrointestinal tumors, or other conditions that the investigator determines may cause gastrointestinal bleeding or perforation or obstruction;
8. History of second primary malignancy within 5 years prior to enrollment, excluding basal cell skin carcinoma or in-situ cervical carcinoma after radical resection;
9. Have known active infection, including but not limited to human immunodeficiency virus (HIV) infection, a history of liver disease known to be significant, including but not limited to hepatitis B virus (HBV) infection and HBV DNA positive (≥1×104/ml); hepatitis C virus infection (HCV) with positive HCV RNA (≥1×103/ml), or cirrhosis, etc.
10. Unresolved toxicities from prior therapy of > grade 1, excluding alopecia; Any other disorders, metabolic abnormality, physical examination abnormality, or laboratory abnormality which has reason to suspect that the patient not suitable for the study or will affect the interpretation of the results. Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-23 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
progression-free survival(PFS) | from the date of randomization up to 36 months
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first,

SECONDARY OUTCOMES:
objective response rate(ORR) | from the date of randomization up to 36 months
  ORR was defined as the percentage of participants who had shown complete response (CR) or partial response (PR) as the best overall response in accordance with the RECIST 1.1 criteria after randomization.
disease control rate(DCR) | from the date of randomization up to 36 months
  Defined as the percentage of patients who have achieved complete response (CR), partial response (PR) and stable disease (SD).
overall survival(OS) | from the date of randomization up to 36 months
  OS was defined as the time from the day of randomization (Day 0) until death by all causes.
Adverse Events(safety) | Up to 28 days after discontinuation of study drug or start of subsequent therapy.
  Adverse events were recorded according to Common Terminology Criteria for Adverse Events (version 5.0) of the National Cancer Institute that participants received at least one dose of protocol treatment after randomization.
Duration of Response (DOR) | from the date of randomization up to 36 months
  From the date of response until the date of first documented disease progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Hao, Dr., Principal Investigator — Qilu hospital of Shandong University, China
Locations (1):
- Qilu hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No